CLINICAL TRIAL: NCT04152018
Title: A PHASE 1 STUDY TO EVALUATE THE SAFETY, PHARMACOKINETICS, AND PHARMACODYNAMICS OF ESCALATING DOSES OF PF-06940434 IN PATIENTS WITH ADVANCED OR METASTATIC SOLID TUMORS
Brief Title: Study of PF-06940434 in Patients With Advanced or Metastatic Solid Tumors.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study termination was based on strategic considerations and not due to specific safety reasons or a request from a regulatory authority.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C3891001; 2020-004009-29 (EudraCT Number)
Record Dates: First submitted 2019-10-30; First posted 2019-11-05 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck; Renal Cell Carcinoma; Ovarian Cancer; Gastric Cancer; Esophageal Cancer; Lung Squamous Cell Carcinoma; Pancreatic Cancer; Bile Duct Cancer; Endometrial Cancer; Melanoma Cancer; Urothelial Cancer
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Renal Cell; Ovarian Neoplasms; Stomach Neoplasms; Esophageal Neoplasms; Pancreatic Neoplasms; Bile Duct Neoplasms; Endometrial Neoplasms | interventions — spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Dose Escalation (Experimental): Single Agent Dose Escalation
  Interventions: Drug: PF-06940434
- Dose Finding Anti-PD-1 Combination 1 (Experimental): Part 1B PF-06940434 plus anti-PD-1
  Interventions: Drug: PF-06940434; Drug: PF-06801591
- Dose Expansion Arm A (Experimental): PF-06940434 with anti-PD-1 in SCCHN
  Interventions: Drug: PF-06940434; Drug: PF-06801591
- Dose Expansion Arm B (Experimental): PF-06940434 with anti-PD-1 in RCC
  Interventions: Drug: PF-06940434; Drug: PF-06801591
- Dose Expansion, Arm C (Experimental): PF-06940434 with anti-PD-1 (both Q3W)
  Interventions: Drug: PF-06940434; Drug: PF-06801591

INTERVENTIONS:
Drug: PF-06940434 — PF-06940434 is given intravenously (IV) every 2 or 4 weeks in a 28 day cycle or every 3 weeks in a 21 day cycle. Multiple dose levels will be evaluated
Drug: PF-06801591 — PF-06801591 will be administered subcutaneously on Day 1 of each 28 day cycle or Day 1 of each 21 day cycle.
  Other Names: Anti-PD-1
  Arms: Dose Expansion Arm A; Dose Expansion Arm B; Dose Expansion, Arm C; Dose Finding Anti-PD-1 Combination 1

SUMMARY:
Open-label, multi-center, non-randomized, multiple dose, safety, tolerability, pharmacokinetic, and pharmacodynamics and clinical activity study of PF-06940434 (Integrin alpha-V/beta-8 Antagonist) in patients with SCCHN (Squamous Cell Carcinoma of the Head and Neck), renal cell carcinoma (RCC - clear cell and papillary), ovarian, gastric, esophageal, esophageal (adeno and squamous), lung squamous cell, pancreatic and biliary duct, endometrial, melanoma and urothelial tumors. This study contains two parts, single agent dose escalation (Part 1A), dose finding of PF 06940434 in combination with anti-PD-1 (Part 1B) and dose expansion (Part 2). Part 2 Dose Combination Expansion will enroll participants into 3 cohorts at doses determined from Part 1B in order to further evaluate the safety of PF-06940434 in combination with anti-PD-1.

ELIGIBILITY:
Inclusion Criteria:

- Histological or cytological diagnosis of SCCHN, RCC (clear cell and papillary cell), ovarian, gastric, esophageal (adeno and squamous), lung squamous cell, pancreatic and biliary duct, endometrial, melanoma, or urothelial cancer.

Part 2:

* Arm A SCCHN:

  * Primary tumor location of the oral cavity, oropharynx, hypopharynx or larynx.
  * PDL-1 expression positive and CPS ≥1. No prior systemic therapy administered in the recurrent or metastatic setting (except for systemic therapy given as part of a multimodal treatment for locally advanced disease).
* Arm B RCC (clear cell):

  * 1 or 2 prior lines of therapy including PD-L1/PD-1 immunotherapy in combination or sequentially with antiangiogenic directed treatment
* Adequate bone marrow, kidney and liver function.
* Performance status of 0 or 1.

Exclusion Criteria:

* Participant disease status is suitable for local therapy administered with curative intent.
* Hypertension that cannot be controlled by medications.
* Active or prior autoimmune disease
* Active, uncontrolled bacterial, fungal, or viral infection, including (but not limited to) Hepatitis B, Hepatitis C, and known Human Immunodeficiency Virus infection or Acquired Immunodeficiency Syndrome-related illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with Dose-limiting toxicities (DLT) for Dose Escalation and Dose Finding | Baseline up to 28 Days (Cycle 1)
Number of Participants With Clinically Significant Change From Baseline in Laboratory Abnormalities | Baseline up to approximately 24 months
Number of Participants With Adverse Events (AEs) According to Severity | Baseline up to approximately 24 months
Number of Participants With Adverse Events (AEs) According to Seriousness | Baseline up to up to approximately 24 months
Number of Participants With Adverse Events (AEs) by Relationship | Baseline up to approximately 24 months
Progression-Free Survival (PFS) for Dose Expansion | Baseline up to 24 Months
  The period from study entry until disease progression, death or date of last contact.
Objective Response Rate - Percentage of Participants With Objective Response in Dose Expansion | Baseline up to 24 months
Duration of Response (DR) for Dose Expansion | Baseline up to 24 Months

SECONDARY OUTCOMES:
PF-06940434 after multiple doses PK parameters (Cmax). | Pre-dose on Cycle 1 Day 1 and on days 3, 8, and 15 of Cycle 1; Day 1 and Day 15 of Cycles 2 and 3; Days 1, 3, 8, and 15 of Cycle 4 and Pre-dose on Day 1 of every cycle thereafter and at end of treatment (each cycle is 28 days).
  Maximum observed plasma concentration of PF-06940434.
Area under the curve from time zero extrapolated to the last quantifiable dose of PF-06940434. | Pre-dose on Cycle 1 Day 1 and on days 3, 8, and 15 of Cycle 1; Day 1 and Day 15 of Cycles 2 and 3; Days 1, 3, 8, and 15 of Cycle 4 and Pre-dose on Day 1 of every cycle thereafter and at end of treatment (each cycle is 28 days).
  Time zero extrapolated to the last quantifiable time point prior to the next dose.
Systemic Clearance (CL) | Pre-dose on Cycle 1 Day 1 and on days 3, 8, and 15 of Cycle 1; Day 1 and Day 15 of Cycles 2 and 3; Days 1, 3, 8, and 15 of Cycle 4 and Pre-dose on Day 1 of every cycle thereafter and at end of treatment (each cycle is 28 days).
  CL is a quantitative measure of the rate at which a drug substance is removed from the body.
Volume of Distribution (Vd) | Pre-dose on Cycle 1 Day 1 and on days 3, 8, and 15 of Cycle 1; Day 1 and Day 15 of Cycles 2 and 3; Days 1, 3, 8, and 15 of Cycle 4 and Pre-dose on Day 1 of every cycle thereafter and at end of treatment (each cycle is 28 days).
Incidence and titers of anti-drug antibodies (ADA) against PF-06940434. | Pre-dose on Days 1 and 15 of Cycle 1, pre-dose on Day 1 of Cycles 2 and 3, pre-dose on Day 1 of Cycle 4, pre-dose on Day 1 of every cycle thereafter and at end of treatment (each cycle is 28 days).
Incidence and titers of neutralizing antibodies (NAb) against PF-06940434. | Pre-dose on Days 1 and 15 of Cycle 1, pre-dose on Day 1 of Cycles 2 and 3, pre-dose on Day 1 of Cycle 4, pre-dose on Day 1 of every cycle thereafter and at end of treatment (each cycle is 28 days).
  Titers of neutralizing antibodies (NAb) against PF-06940434.
PK parameters of PF-06940434 and PF-06801591 (Cmax). | Pre-dose on Cycle 1 Day 1 and on day 15 of Cycle 1; Day 1 of Cycles 2 and 3; Days 1, 3, 8, and 15 of Cycle 4 and Pre-dose on Day 1 of every cycle thereafter and at end of treatment (each cycle is 28 days)
  Maximum observed plasma concentration after multiple doses of PF-06940434 and PD-1 (PF-06801591).
Area under the curve from time zero extrapolated to the last quantifiable dose of PF-06940434 and PF-06801591. | Pre-dose on Cycle 1 Day 1 and on day 15 of Cycle 1; Day 1 of Cycles 2 and 3; Days 1, 3, 8, and 15 of Cycle 4 and Pre-dose on Day 1 of every cycle thereafter and at end of treatment (each cycle is 28 days)
  Area under the curve from time zero extrapolated to the last quantifiable dose of PF-06940434 and PF-06801591.
Characterize the multiple dose PK of PF-06940434 following intravenous administration in combination with PF-06801591. | Cycle 4 Day 1 (each cycle is 28 days)
  Maximum observed plasma concentration of PF-06940434.
Area under the curve from time zero extrapolated to the last quantifiable dose of PF-06940434. | Cycle 4 Day 1 (each cycle is 28 days)
  Time zero extrapolated to the last quantifiable time point prior to the next dose.
Number of participants with increased T-cells after PF-06940434 treatment. | Pre-dose on Day 1 of Cycle 1; pre-dose on Day 1 of Cycles 2 and 3 (each cycle is 28 days)
Progression-Free Survival (PFS) for Dose Expansion | Baseline to measured progression (up to approximately 24 months)
  The period from study entry until disease progression, death or date of last contact.
Duration of Response (DR) | Baseline up to approximately 24 Months
Number of Participants With Objective Response for Dose Expansion portion | Baseline up to 24 months
Disease Control Rate (DCR) | Every 8 weeks from the time of enrollment up to 2 years
  DCR is defined as the percent of participants with a confirmed complete response (CR), partial response (PR) or stable disease (SD) according to RECIST 1.1.
Trough concentrations of PF-06940434 and PF-06801591 in Dose Expansion | Day 1 of Cycle 1 though 4, Day 1 of every 2 Cycles starting from Cycle 5 up to 24 months (each cycle is 28 days). For Part 2 Cohort 3, Day 1 of Every Cycle (each cycle is 21 days)
Plasma Decay Half-Life (t1/2) | Pre-dose on Cycle 1 Day 1 and on days 3, 8, and 15 of Cycle 1; Day 1 and Day 15 of Cycles 2 and 3; Days 1, 3, 8, and 15 of Cycle 4 and Pre-dose on Day 1 of every cycle thereafter and at end of treatment (up to 24 Months) [each cycle is 28 days]
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Incidence and titers of anti-drug antibodies (ADA) against PF-06801591 in Dose Finding and Dose Expansion | Pre-dose on Days 1 and 15 of Cycle 1, pre-dose on Day 1 of Cycles 2 and 3, pre-dose on Day 1 of Cycle 4, pre-dose on Day 1 of every cycle thereafter and at end of treatment (up to 24 Months) [each cycle is 28 days].
  Incidence and titers of anti-drug antibodies (ADA) against PF-06801591.
Incidence and titers of neutralizing antibodies (NAb) against PF-06801591 in Dose Finding and Dose Expansion. | Pre-dose on Days 1 and 15 of Cycle 1, pre-dose on Day 1 of Cycles 2 and 3, pre-dose on Day 1 of Cycle 4, pre-dose on Day 1 of every cycle thereafter and at end of treatment (up to 24 Months) [each cycle is 28 days].
  Incidence and titers of neutralizing antibodies (NAb) against PF-06801591.
Overall Survival | From baseline to up to 2 years after last dose of study drug
  The period from study entry until death or date of last contact (24 months)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (31):
- United States (18):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - HonorHealth Scottsdale Shea Medical Center, Scottsdale, Arizona
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - UCLA Hematology Oncology, Los Angeles, California
  - UCLA Hematology/Oncology, Santa Monica, California
  - Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Siteman Cancer Center - St. Peters, City of Saint Peters, Missouri
  - Siteman Cancer Center - West County, Creve Coeur, Missouri
  - Siteman Cancer Center - North County, Florissant, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University School of Medicine Siteman Cancer Center, St Louis, Missouri
  - Siteman Cancer Center - South County, St Louis, Missouri
  - Duke Univ. Medical Center/Duke Cancer Center, Durham, North Carolina
  - Investigational Chemotherapy Service, Durham, North Carolina
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology, San Antonio, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
- Southern Medical Day Care Centre, Wollongong, New South Wales, Australia
- Slovakia (7):
  - Onkologicky ustav sv. Alzbety, s.r.o., Bratislava
  - Univerzitna nemocnica Bratislava, Bratislava
  - Narodny ustav srdcovych a cievnych chorob, a.s., Bratislava
  - MR Poprad s.r.o., Komárno
  - KARDIO, s.r.o., Poprad
  - POKO Poprad, s.r.o., Ambulancia klinickej onkologie, Poprad
  - Nemocnica Poprad a.s., Poprad
- South Korea (2):
  - Asan Medical Center, Seoul, Seoul-teukbyeolsi [seoul]
  - Severance Hospital, Yonsei University Health System, Seoul
- Taiwan (3):
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3891001